CLINICAL TRIAL: NCT00707018
Title: Immobilization in External Rotation After First Time Anterior Shoulder Dislocation: A Prospective Randomized Study
Brief Title: Immobilization in External Rotation After First Time Anterior Shoulder Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0088
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External rotation shoulder sling (Experimental): External rotation shoulder sling
  Interventions: Device: External rotation shoulder sling
- Internal rotation shoulder sling (Active Comparator): Internal rotation shoulder sling
  Interventions: Device: Internal rotation shoulder sling

INTERVENTIONS:
Device: External rotation shoulder sling — The external rotation sling will be adjusted to position the injured upper extremity in 90 degrees of elbow flexion, 0 degrees of shoulder abduction and flexion, and 10 to 15 degrees of external rotation at the shoulder.
  Arms: External rotation shoulder sling
Device: Internal rotation shoulder sling — The internal rotation sling will be adjusted to position the injured upper extremity in 90 degrees of elbow flexion, 0 degrees of shoulder abduction and flexion, and 70 to 80 degrees of internal rotation at the shoulder.
  Arms: Internal rotation shoulder sling

SUMMARY:
Comparison of immobilization in internal versus external rotation after first time anterior shoulder dislocation.

DETAILED DESCRIPTION:
The purpose of this study is to compare immobilization in internal versus external rotation after first time anterior shoulder dislocation, and thereby increase our knowledge about the best standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 30 years of age
* Willing to participate in follow-up for at least two years
* Acute, first-time, traumatic, isolated anterior dislocation of the shoulder

Exclusion Criteria:

* Previous instability of the affected shoulder
* A history of significant ligamentous laxity or demonstrated multi-directional instability of the opposite shoulder
* Inability or unwillingness to comply with sling immobilization, rehabilitative protocol, or required follow-up assessments
* Incompetent or unwilling to consent
* A medical condition making the patient unable to wear a sling
* Significant associated fracture (Exception Hill Sachs of >20% or bony Bankart lesions>10%)
* Neurovascular compromise of the affected limb
* Concomitant ipsilateral upper extremity injuries which may affect the patient's ability to participate in, or benefit from, a rehabilitative program.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2004-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Recurrent instability consisting of a documented episode of anterior shoulder dislocation or multiple episodes of shoulder subluxation. | 24 months

SECONDARY OUTCOMES:
Patient self reported outcome measures | 24 Months
Time to return to work or sport | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Eric C McCarty, MD, Principal Investigator — University of Colorado, Denver
Locations (8):
- United States (8):
  - CU Sports Medicine, Boulder, Colorado
  - St. Anthony Hospitals, Winter Park, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of New Mexico, Albuquerque, New Mexico
  - Summa Healthcare, Akron, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Inland Orthopaedics, Pullman, Washington